CLINICAL TRIAL: NCT06215092
Title: Perinatal, Cognitive and Social-emotional Correlates of Neurodevelopmental Disorders and Learning Difficulties in Children and Adolescents, From a Biopsychosocial Perspective.
Brief Title: Perinatal and Psychological Correlates of Neurodevelopmental Disorders in Children.
Status: Completed | Type: Observational
Sponsor: Bartosz M. Radtke (Other Government)
Responsible Party: Sponsor-Investigator, Bartosz M. Radtke, PhD, Laboratory of Psychological and Educational Tests
Organization: Laboratory of Psychological and Educational Tests (Other Government)
Other Study IDs: 2023/PTPiP/1
Record Dates: First submitted 2024-01-10; First posted 2024-01-22 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Perinatal Condition; Neurodevelopmental Disorders; Social Functioning; Child Development; Adolescent Development
Keywords: hypoxia; dyslexia; mild intellectual disability; ADHD; ASD; Learning difficulties; social-emotional functioning
MeSH Terms: conditions — Neurodevelopmental Disorders; Social Adjustment; Hypoxia; Dyslexia; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Developmental learning disorder: Children above 5 years old, with formal diagnosis of Developmental learning disorder.
  Interventions: Other: Psychological assessment
- Disorder of intellectual development, mild: Children above 5 years old, with formal diagnosis of Disorder of intellectual development, mild.
  Interventions: Other: Psychological assessment
- Attention deficit hyperactivity disorder: Children above 5 years old, with formal diagnosis of Attention deficit hyperactivity disorder (ADHD).
  Interventions: Other: Psychological assessment
- Autism spectrum disorder: Children above 5 years old, with formal diagnosis of Autism spectrum disorder (ASD).
  Interventions: Other: Psychological assessment
- Learning difficulties: Children above 5 years old, with difficulties in reading and/or writing without formal diagnosis of Developmental learning disorder.
  Interventions: Other: Psychological assessment
- Control group: Children above 5 years old without formal diagnosis of neurodevelopmental disorders.
  Interventions: Other: Psychological assessment

INTERVENTIONS:
Other: Psychological assessment — Psychological assessment of cognitive and social-emotional functioning.

SUMMARY:
The goal of this observational study is to investigate perinatal, cognitive and social-emotional correlates of neurodevelopmental disorders and educational difficulties in children and adolescents.

The study group consist of minimal 500 childrens over 5 years of age who will be examined by qualified diagnosticians. Participants will be evaluated with tasks related to the studied variables: cognitive functioning, social-emotional functioning. Furthermore informations regarding social-emotional functioning of children, will be collected from parents and teachers.

The main questions it aims to answer are:

1. Is there a relationship between perinatal factors and the risk of occurrence of neurodevelopmental disorders and/or learning difficulties?
2. Is there a specific pattern of cognitive functioning in children and adolescents with indicated neurodevelopmental disorders and/or learning difficulties?
3. Is there a specific pattern of social-emotional functioning in children and adolescents with indicated neurodevelopmental disorders and/or learning difficulties?
4. Do gender and age moderates specific patterns of cognitive and social-emotional functioning in the studied groups?

Researchers will compare the following groups of children over 5 years old:

1. With perinatal risks factors
2. With neurodevelopmental disorders:

   1. Developmental learning disorder
   2. Disorder of intellectual development, mild
   3. Attention deficit hyperactivity disorder
   4. Autism spectrum disorder
3. With Learning difficulties
4. Control group

ELIGIBILITY:
Inclusion criteria for neurodevelopmental disorder groups:

* age between 5 to 18 y.o.
* diagnosed neurodevelopmental disorders, depending on the study group: 1) Developmental learning disorder; 2) Disorder of intellectual development, mild; 3) Attention deficit hyperactivity disorder; 4) Autism spectrum disorder

Inclusion criteria for learning difficulties:

* age between 5 to 18 y.o.
* difficulty in reading and/or writing without a diagnosis of Developmental learning disorder

Inclusion criteria for control group

* age between 5 to 18 y.o.
* without a diagnosis of any neurodevelopmental disorder

Exclusion criteria for learning difficulties

- diagnosis of Developmental learning disorder

Exclusion criteria for all groups:

* age below 5 y.o. and equal to or above 19 y.o.
* diagnosis of any neurodevelopmental disorders

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Polish children and adolescents attending to formal education schools in age 5 to 18 years old.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-11-20 (Actual); Study Completion 2025-12-19 (Actual)

PRIMARY OUTCOMES:
Perinatal risks factors | Data collected immediately after childbirth.
  Data from medical documentations including: birth weight, body length, head and chest circumference, Apgar score, interventions supporting breathing and blood circulation.
Memory and learning | Juli 1, 2022 until April 30, 2024
  Test of Memory and Learning (second edition). A standardized test measuring memory functioning and learning abilities in children and adolescents. The test includes four basic factors (Verbal Memory, Nonverbal Memory, Complex Memory, and Delayed Recall) and five supplementary factors (Attention/Concentration, Sequential Memory, Free Recall, Associative Recall and Learning).
Cognitive abilities | Juli 1, 2022 until April 30, 2024
  Specialized Learning Disabilities Battery. A standardized test allowing the assessment of cognitive processes important in learning and selected school skills in children and adolescents. The test consists of six scales and fifteen subscales: 1) Visuospatial Processing (Analysis and Synthesis, Rotation Rate, Visual Memory); 2) Auditory-Linguistic Processing (Phonetic Coding - Linguistic Aspect, Phonetic Coding - Cognitive Complexity, Resistance to Distractors); 3) Reading and Writing (Decoding, Comprehension, Writing, Spelling); 4) Long-term Memory (Associative Memory, Memory of Meanings); 5) Knowledge (General Knowledge, Lexical Knowledge); 6) Processing Rate (Speed of Perception).
Social-emotional competence | Juli 1, 2022 until April 30, 2024
  The Social-Emotional Evaluation (SEE). A standardized test designed to evaluate aspects of emotional and social awareness, wich are part of the social-emotional competence. The SEE contains four core subtests, one supplemental subtest, and a Social Emotional Questionnaire: 1) Identifying Common Emotions; 2) Identifying Emotional Reactions; 3) Understanding Social Gaffes; 4) Understanding Conflicting Messages; Supplemental Subtest: Recognizing Facial Expressions; The Social Emotional Questionnaire assesses general social-emotional intelligence, based on both a parent/caregiver and an educator/specialist responds.
Socio-demographic data | Juli 1, 2022 until April 30, 2024
  Authors survey of socio-demographic data, including: gender, month and year of birth, size of place of residence, region of residence, school, class, age of starting education, average grade from the last semester, diagnosis (if any), parents education level

SECONDARY OUTCOMES:
General intellectual functioning | Juli 1, 2022 until April 30, 2024
  Stanford-Binet Intelligence Scales-Fifth Edition (SB5). A standardized test which assessment two main intellectual domain (Nonverbal and Verbal). Each domain consist of five scales (Fluid Reasoning, Knowledge, Quantitative Reasoning, Visual-Spatial Processing, and Working Memory). This test is based on the Cattel-Horn-Carroll Intelligence Theory (CHC).
Nonverbal intellectual functioning | Juli 1, 2022 until April 30, 2024
  Test of Nonverbal Intelligence-Fourth Edition (TONI-4). A norm-referenced instrument that measures a General Intelligence. The TONI-4 has two equivalent forms: Form A and Form B. Each form consists of 60 items, all of which are abstract/figural.
Executive functions | Juli 1, 2022 until April 30, 2024
  Nonverbal Stroop Card Sorting Test (NSCST). A standardized, nonverbal Stroop test for cognitive-process, executive functioning and neuropsychological assessment. Test contain two groups of cards, which examinee have to sort cards according to presented visual stimulus. Additionally, the test includes an observational scale that allows to assessed the following processes: attention, impulse control, level of activity, anxiety and reactivity.
Learning difficulties | Juli 1, 2022 until April 30, 2024
  The Battery for Assessment of the Causes of Learning Difficulties. A set of tests to assess the occurrence of developmental learning disorders of reading and writing in school-age children. The battery consists of tests diagnosing: visual-spatial Functions (visual-spatial perception and speed of visual perception when working with visual material, eye-hand coordination, structuring of perception, attention and visual-motor control when working with complex material and short-term visual memory capacity), auditory-linguistic functions (phoneme hearing, phonological memory, ability to perform sound-phoneme analysis, sound abstraction and synthesizing sounds, attention and phonological memory), perceptual-motor integration, reading and writing skills.
Communication, social interaction, restricted and repetitive behaviors | Juli 1, 2022 until April 30, 2024
  The Autism Diagnostic Observation Schedule, Second Edition (ADOS-2). A tool consisting of a set of tests and standardized components that allow to observe the person being examined during a naturally occurring interaction with a diagnostician. It consists of five Modules intended for respondents of different ages and levels of development of linguistic expression. ADOS-2 allows to assess various aspects of behavior, representing five categories: Language and communication, Social interactions, Play/Imagination, Stereotypical behavior and Rigid interests, Other behaviors that differ from the norm. The obtained data are analyzed on two scales: Social Affect and Restricted and Repetitive Behavior, as well as a total score allowing to assess the occurrence and level of severity of Autism spectrum disorder.
Early social-emotional development | Juli 1, 2022 until April 30, 2024
  The Emotional Development Scale for Children Aged 3-6. A standardized test for assessing the emotional development of preschool children, which consists of three diagnostic scales: 1) Recognizing emotions, 2) Naming emotions and 3) Emotions in social situations.
Social-emotional development | Juli 1, 2022 until April 30, 2024
  A part of Intelligence and Development Scales - 2nd edition (IDS-2), assessing social-emotional skills in a school-aged children. A standardized test consisting of three diagnostic scales: 1) Recognizing Emotions, 2) Regulating Emotions, 3) Social Strategies.

CONTACTS AND LOCATIONS:
Overall Officials: Urszula Sajewicz-Radtke, Ph.D., Principal Investigator — Laboratory of Psychological and Educational Tests; Bartosz M Radtke, Ph.D., Study Director — Laboratory of Psychological and Educational Tests; Ariadna Łada-Maśko, Ph.D., Principal Investigator — Laboratory of Psychological and Educational Tests
Locations (1):
- Laboratory of Psychological and Educational Tests, Gdansk, Pomeranian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sajewicz-Radtke U, Radtke BM, Jurek P, Olech M, Lada-Masko A. Beyond Uniform Impairment: Investigating Declarative Memory Profiles in Nonspecific Mild Intellectual Disability Using Latent Profile Analysis. J Intellect Disabil Res. 2025 Dec;69(12):1425-1434. doi: 10.1111/jir.70039. Epub 2025 Sep 3. PMID 40903989